CLINICAL TRIAL: NCT02183740
Title: Effect of an Educational Program for Staff in Nursing Homes Concerning Patients Fecal Incontinence: a Cluster-randomized Controlled Trial
Brief Title: Effect of an Educational Program for Staff in Nursing Homes Concerning Patients Fecal Incontinence
Acronym: EPSPFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Nurses Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HiST05
Record Dates: First submitted 2014-06-26; First posted 2014-07-08 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Fecal Incontinence
Keywords: Education; Nurses; Nursing homes; Fecal incontinence; Cluster-randomized controlled trial
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multifaceted educational program (Experimental): A multifaceted educational program for nursing home staff consisting of:
  1. One seven hours educational meeting (interactive workshop) conducted in the nursing home. Theoretical input and case-base discussions considering guidelines for nurse led assessment og interventions of patients fecal incontinence.The content will be made available as educational material.
  2. Recruitment of one local opinion leader per nursing home unit.
  3. Seven educational outreach meetings (1 hour 30 minutes per meeting) during the three months intervention period.
  Interventions: Behavioral: Multifaceted educational program
- Control (No Intervention): The control arm will not receive any educational program and will continue with usual care. Data with information about ordinary care will be gathered as part of the data collection procedure in the study.

INTERVENTIONS:
Behavioral: Multifaceted educational program
  Arms: Multifaceted educational program

SUMMARY:
Fecal incontinence (FI) has an increasing prevalence in the geriatric population which cannot be explained by co-morbidity or anatomical and psychological changes of aging alone. In the nursing home population previous studies suggest a prevalence between 10 and 69%, but is most often reported to be between 40 and 55%. FI leads to a high direct and indirect economic burden to the health-care system, and is an important cause og institutionalization of the elderly patients. In addition, FI is associated with shame, social isolation and reduced quality of life.

The importance of identifying treatable causes of FI in the frail elderly, rather than just managing passively, is strongly emphasized. It is indicated that the level of awareness among health personnel regarding appropriate assessment and treatment options is limited, and that FI is considered a normal part of aging.

This study is based on the assumption that FI among nursing home patients can be prevented, cured or ameliorated by offering nursing home staff knowledge of best practise. The primary objective of the study is to test the hypothesis that a multifaceted educational program for staff on assessment and treatment of FI, is associated with a reduction in patients' frequency of FI.

The design of the study is a two armed cluster randomized trail (C-RCT) with a repeated cross-sectional approach.The results will be analysed according to multilevel and longitudinal modelling, and the study will use mixed effect models with the cluster treated as a random effect.

ELIGIBILITY:
Inclusion Criteria:

Nursing homes with similar:

* patients characteristcs
* care staff/patients ratio
* general practitioner consultancy

Patients:

- All patients on long term care residency (residency >month)

Registered Nurses/authorized social educators:

- All working half time or more

Exclusion Criteria:

Nursing homes:

- With some kind of speciality (eks rehabilitation, dementia)

Patients:

- Short term care residency

Registered nurses/authorized social educator:

* Working less than half time
* Working only night shifts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in frequency of fecal incontinence among patients | Baseline, after 3 months and after 6 months
  As measured by The Long-Term Care Facilities Assessment System (interRAI-LTCF 2012), section H: Continence. Because of relatively high risk of death and movement out of clusters, a repeated cross-sectional opproach to analyses will be used. Frequency of FI will thereby be analysed on a across-sectional group level.

SECONDARY OUTCOMES:
Remission of fecal incontinence among patients | Baseline, after 3 months and after 6 months
  For remission of FI a cohort approach to data analyses with only those identified with FI at baseline and still present at 3 and 6 month follow-up, will be included in the analyses
Change in knowledge among registered nurses and authorized social educators | Baseline, after 3 months and after 6 months
  Measured my a multiple choice test
Change in FI-related concerns among patients | Baseline, after 3 months and after 6 months
  Relevant concerns as measured by The Long-Term Care Facilities Assessment System (interRAI-LTCF 2012) are: Mood and behavior, psycho-social wellbeing, urinary continence, constipation, diarrhea, skin condition, participation in activities
Correlates of FI among patients | Baseline, after 3 months and after 6 months
  Relevant correlates as measured by The Long-Term Care Facilities Assessment System (interRAI-LTCF 2012) are: cognitive functioning, communication and vision, functionality and mobility, medical diagnosis, mouth and nutrition status, medications, treatment, examination/procedures
Change in behavior among health personnel | Baseline, after 3 months and after 6 months
  Measured by analyses of patient assessments and interventions as documented by health personnel in the electronic patient record and by the Fecal Incontinence in Nursing Home Patients questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anne G Vinsnes, Professor, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Sor Trondelag University College, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blekken LE, Vinsnes AG, Gjeilo KH, Morkved S, Salvesen O, Norton C, Nakrem S. Effect of a multifaceted educational program for care staff concerning fecal incontinence in nursing home patients: study protocol of a cluster randomized controlled trial. Trials. 2015 Mar 1;16:69. doi: 10.1186/s13063-015-0595-3. PMID 25887238
- [Background] Blekken LE, Nakrem S, Gjeilo KH, Norton C, Morkved S, Vinsnes AG. Feasibility, acceptability, and adherence of two educational programs for care staff concerning nursing home patients' fecal incontinence: a pilot study preceding a cluster-randomized controlled trial. Implement Sci. 2015 May 23;10:72. doi: 10.1186/s13012-015-0263-8. PMID 26002520